CLINICAL TRIAL: NCT02004457
Title: Engaging HIV Patients in Primary Care by Promoting Acceptance
Acronym: HIV Engage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Butler Hospital (Other)
Collaborators: Brown University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R34MH098694-02 (NIH)
Record Dates: First submitted 2013-11-26; First posted 2013-12-09 (Estimated); Last update posted 2017-03-09 (Actual); Status verified 2017-03

CONDITIONS: HIV
Keywords: HIV; Primary care; Engagement; Acceptance; Disclosure; Stigma
MeSH Terms: conditions — Social Stigma

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acceptance-based behavior therapy (ABBT) (Experimental): ABBT will consist of 2 sessions. The first session will be used to introduce the concept of acceptance and its possible benefits in the context of life values and patient-identified barriers to care engagement. Following a discussion of life values will be a discussion of which, if any, of these values are currently misaligned with the participant's HIV self-care. At the second session, acceptance-based coping skills will be practiced and a behavioral plan will be developed to targets barriers identified in the first session. These discussions will help the participant clarify how best to align their values with decisions on how to manage his/her HIV (e.g. when and how to disclose, what to expect at appointments).
  Interventions: Behavioral: ABBT
- Treatment-as-usual (TAU) (Placebo Comparator): TAU will consist of the standard sessions all individuals receive as they enter HIV care and attend their first follow-up visit to review lab results. TAU includes identification of environmental barriers to care, assessment of needs for additional care and corresponding referrals (i.e., for depression, substance abuse), and recommendations to attend HIV support groups.
  Interventions: Other: TAU

INTERVENTIONS:
Behavioral: ABBT
  Arms: Acceptance-based behavior therapy (ABBT)
Other: TAU
  Arms: Treatment-as-usual (TAU)

SUMMARY:
Engagement in primary care for People Living with HIV/AIDS (PLWHA) is a significant public health concern because reduced commitment to care puts PLWHA at risk for illness progression, death, and transmission of HIV to others. This project will develop a novel treatment, brief acceptance-based behavior therapy (ABBT), to promote self-acceptance of HIV status as a pathway to reducing engagement barriers. The clinical and public health impact of this project will be the development of a simple, low-cost, disseminable intervention that enhances longitudinal commitment to care so PLWHA can obtain effective medical treatments that will prolong survival and improve quality of life. We hypothesize that individuals randomized to brief ABBT will showed increased longitudinal attendance of primary care appointments.

ELIGIBILITY:
Inclusion Criteria:

* new to the primary care clinic
* HIV+
* between 18 and 60 years old
* entering HIV care for the first time
* able to speak and read English sufficiently to be able to complete the study procedures
* have access to a telephone

Exclusion Criteria:

* psychiatrically or cognitively impaired

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2013-03; Primary Completion 2016-05 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Frequency of attended primary care medical appointments | 9 months
  The number of primary care medical appointments a participant attends over the course of 9 months.
Acceptance and Action Questionnaire-2 | 9 months
  A modified version of the Acceptance and Action Questionnaire-2 (AAQ-2) will be used to quantify the degree to which participants accept their HIV diagnosis and related stresses.
HIV Disclosure Scale | 9 months
  The HIV Disclosure Scale will be used to quantify how willing participants are to disclose their HIV status to others.

SECONDARY OUTCOMES:
Berger HIV Stigma Scale | 9 months
  The Berger HIV Stigma Scale will used to measure the degree to which participants experience HIV-related stigma.
Disclosure to others | 9 months
  The number of individuals to whom the participant discloses his/her HIV status to.
Social Support Questionnaire | 9 months
  The Social Support Questionnaire will be used to measure participants' perceived social support.

CONTACTS AND LOCATIONS:
Locations (1):
- Butler Hospital, Providence, Rhode Island, United States

REFERENCES:
- [Derived] Moitra E, LaPlante A, Armstrong ML, Chan PA, Stein MD. Pilot Randomized Controlled Trial of Acceptance-Based Behavior Therapy to Promote HIV Acceptance, HIV Disclosure, and Retention in Medical Care. AIDS Behav. 2017 Sep;21(9):2641-2649. doi: 10.1007/s10461-017-1780-z. PMID 28451891